CLINICAL TRIAL: NCT06184971
Title: Biliary Atresia Research Network Northeast (BARNN)
Brief Title: Biliary Atresia Research Network Northeast
Acronym: BARNN
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 2000035645; 000 (Other: CTGTY)
Record Dates: First submitted 2023-12-13; First posted 2023-12-29 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Biliary Atresia
MeSH Terms: conditions — Biliary Atresia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi-center retrospective chart review to compile a data repository of the management and outcomes of children with biliary atresia. Overall, investigators aim to evaluate which specific factors contribute to improved patient outcomes, to help guide potential improvements in patient care and resource utilization.

DETAILED DESCRIPTION:
Biliary atresia is quite rare, with only 0.73 cases per 10,000 births in the US. Due to this rarity and the geographical spread of the US, the small number of cases end up being dispersed amongst the various pediatric hospitals, which leads to certain hospitals only encountering an affected patient once per decade. This rarity and dispersion makes biliary atresia difficult for researchers to study: single-institution studies are limited by low power and only provide narrow snapshots, whereas large NIH-sponsored consortia report highly selected outcomes from only the largest or most dedicated centers and have largely excluded New England. This leaves a significant knowledge gap regarding the management and outcomes at more typical hospitals. The purpose of this study is to collect clinical data from all children with biliary atresia at all hospitals providing pediatric surgical care in the Northeast, even very-low-volume hospitals. This is a retrospective study, only involving chart review. There will be no interaction with subjects, intervention, or collection of specimens for the purposes of this study. The data will only include clinical information that was recorded during the normal course of patient care. The subjects will be de-identified before entry into a HIPAA-compliant data repository. This data repository will allow researchers to pool data, to yield adequate statistical power and assess differences in management and outcomes regarding this very rare condition.

ELIGIBILITY:
Inclusion Criteria:

* Children with a healthcare encounter related to biliary atresia at a participating institution during the study period (January 1st, 2012 through December 31st, 2021)
* Age 12 years and younger at the time of the qualifying encounter during the study period (encompassing patients born between January 2nd, 1999 through December 31st, 2021)
* Diagnosis of biliary atresia, based on one of the following ICD-10 codes:

  * Q44.2 Atresia of bile ducts
  * Q44.3 Congenital stenosis and stricture of bile ducts
  * Q44.4 Disorders of the biliary tract with major complication or comorbidity
  * Q44.5 Other congenital malformations of the bile ducts
  * Q44.6 Disorders of the biliary tract without major complication or comorbidity

Exclusion Criteria:

* Patients aged 13 years old or older during the study period (i.e. those born before January 2nd, 1999)
* Patients born and/or diagnosed with biliary atresia after the end of the study period (i.e. those born after December 31st, 2021)
* No diagnosis of biliary atresia
* History of biliary atresia without any episodes of care related to biliary atresia during the study period (e.g. a teenager with history of BA who underwent Kasai procedure as an infant and has no current issues related to their BA and is receiving care for an unrelated reason)

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 12 years and younger (at the time of the qualifying encounter for care) who were diagnosed with biliary atresia, underwent surgical intervention for biliary atresia, and/or had an encounter for care related to biliary atresia at a participating institution during the study period. Patients who did not undergo surgery will be included (e.g. patients who died before surgery).
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Death | 10 years
  Patient death
Kasai procedure | 10 years
  Need for biliary diversion procedure, including the Kasai portoenterostomy
Liver transplant | 10 years
  Need for liver transplant

SECONDARY OUTCOMES:
Clearance of jaundice | 6 months
  Normalization of serum bilirubin after Kasai procedure
Bilirubin level | 10 years
  Serum bilirubin level
Cholangitis | 10 years
  Clinical diagnosis of cholangitis
Bleeding | 10 years
  Post-operative bleeding requiring transfusion or return to the OR
Presentation to ED | 10 years
  Patient presentation to the ED for complication related to biliary atresia
Age at follow-up with providers | 10 years
  Frequency and age at most recent follow-up with Pediatric Surgeon and/or Hepatologist

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cowles, MD, Principal Investigator — Yale University
Locations (14):
- United States (14):
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Medical Center, Portland, Maine
  - Massachusetts General Hospital for Children, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Baystate, Springfield, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Albany Medical Center/Bernard & Millie Duke's Children's Hospital, Albany, New York
  - John R. Oishei Children's Hospital, Buffalo, New York
  - University of Rochester Medical Center/Golisano Children's Hospital, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Rhode Island Hospital/Hasbro Children's Hospital, Providence, Rhode Island